CLINICAL TRIAL: NCT00558363
Title: A Randomised, Double-Blind, Placebo-Controlled Trial Assessing the Efficacy and Safety of Dutasteride (AVODART™) 0.5 mg in Extending the Time to PSA Doubling in Men With Prostate Cancer and Biochemical Failure (PSA Increase) After Radical Therapy With Curative Intent
Brief Title: ARTS - AVODART After Radical Therapy For Prostate Cancer Study
Acronym: ARTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI109924
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2011-12

CONDITIONS: Neoplasms, Prostate; Prostate Cancer After a Radical Treatment
Keywords: Prostate Cancer; AVODART; PSA; dutasteride; PSADT; Prostate specific antigen; radical therapy; doubling time
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avodart (Experimental): Patients will receive a 3-month supply of study drug or placebo. Patients will be instructed to take one capsule by mouth once daily. Study medication will be supplied at 3-month intervals during scheduled clinic visits for a total of 24 months.
  Interventions: Drug: Avodart
- Placebo Arm (Placebo Comparator): Patients will receive a 3-month supply of study drug or placebo. Patients will be instructed to take one capsule by mouth once daily. Study medication will be supplied at 3-month intervals during scheduled clinic visits for a total of 24 months.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Avodart — 0.5 mg administered orally once daily
  Other Names: Avodart/placebo
  Arms: Avodart
Other: placebo — Patients will be randomized at Visit 2 in 1:1 ratio to receive either 0.5 mg dutasteride or placebo
  Arms: Placebo Arm

SUMMARY:
ARI109924 will be a 2-year, multicentre, randomised, double-blind, placebo-controlled trial assessing the efficacy and safety of dutasteride in extending time to prostate specific antigen (PSA) doubling in men who have been treated for clinically localised prostate cancer (PCa) with a radical therapy (radical prostatectomy, primary radiotherapy or salvage radiotherapy) with curative intent but who experience a biochemical failure (PSA rise) afterwards without signs or symptoms of metastases.

DETAILED DESCRIPTION:
A Randomised, Double-Blind, Placebo-Controlled Trial Assessing the Efficacy and Safety of Dutasteride (AVODART™) 0.5 mg in Extending the Time to PSA Doubling in Men with Prostate Cancer and Biochemical Failure (PSA increase) after Radical Therapy with Curative Intent (ARTS - AVODART after Radical Therapy for prostate cancer Study)

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for enrolment in the study must meet all of the following criteria:

* Males <85 years of age
* No clinically relevant abnormal findings on the screening ECG
* Patients with asymptomatic PSA failure following radical therapy with curative intent for clinically localised prostate cancer. PSA failure is defined as:
* After primary radiotherapy:
* 3 rises in PSA levels from nadir PSA, with each determination at least 4 weeks apart and a final PSA level ≥2 ng/mL above nadir PSA
* Time from radiotherapy should be at least 1 year from termination of radiotherapy treatment
* After radical prostatectomy with or without salvage radiotherapy:
* 3 rises in PSA level from nadir PSA, with each determination at least 4 weeks apart and each PSA level ≥0.2 ng/mL and a final PSA level ≥0.4 ng/mL (nadir PSA is defined as the lowest PSA value achieved after therapy)
* Serum PSA levels:
* ≥2 ng/mL and ≤20ng/mL for primary radiotherapy patients
* ≥0.4 ng/ml and ≤10ng/ml for radical prostatectomy with or without salvage radiotherapy patients
* PSADT >3 months and ≤24 months
* Clinical stage T1-T3a N0 M0
* Non-metastatic prostate cancer, as confirmed on a negative bone scan performed within 6 months prior to randomisation (Visit 2)3.
* No evidence of local recurrence in radical prostatectomy or salvage radiotherapy patients
* Expected survival ≥2 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2 (see Appendix 1)

Miscellaneous:

* Able to swallow and retain oral medication
* Able and willing to participate in the full 2 years of the study
* Able to read and write (the MAX-PC questionnaire is self-administered), understand instructions related to study procedures and give written informed consent
* In France, a patient will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Any unstable serious co-existing medical condition(s) including but not limited to myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure or cerebrovascular accident within 6 months prior to Visit 1, or uncontrolled diabetes or peptic ulcer disease which is uncontrolled by medical management
* Abnormal liver function tests (greater than 2 times the upper limit of normal [ULN] for alanine aminotransferase [ALT], aspartate aminotransferase [AST] or alkaline phosphatase [ALP] or >1.5 x ULN for bilirubin).
* Serum creatinine >1.5 x ULN
* History of another malignancy within 5 years that could affect the diagnosis of prostate cancer
* History or current evidence of drug or alcohol abuse within 12 months prior to Visit 1
* History of any illness (including psychiatric) that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient
* Known hypersensitivity to any 5-AR inhibitor or to any drug chemically related to dutasteride

Disease characteristics:

* Serum PSA levels
* >20 ng/mL in primary radiotherapy patients
* >10 ng/mL in radical prostatectomy with or without salvage radiotherapy patients
* PSADT ≤3 months or >24 months
* Biochemical failures in post brachytherapy patients
* Clinical stage N+ or M+
* Patient has previously been treated for prostate cancer with any of the following:
* Chemotherapy
* Oestrogens (e.g. megestrol, medroxyprogesterone, cyproterone, Diethylstilbestrol [DES])
* Drugs with anti-androgenic properties (e.g. spironolactone if >50mg/day, flutamide, bicalutamide, ketoconazole, progestational agents), (except when used for adjuvancy or neoadjuvancy in the context of a primary radical treatment in which case their use should have been for no more than 6 months and should have completed at least 1 year before Visit 1 [Note: the use of topical ketoconazole is permitted prior to and during the study and the use of cimetidine is permitted prior to study entry]
* GnRH analogues (e.g., leuprolide, goserelin) except when used for adjuvancy or neoadjuvancy in the context of a primary radical treatment (in this case use should have been for no more than 6 months and should have finalised at least 1 year before Visit 1)
* Orchiectomy

Concomitant medications:

* Glucocorticoids, except inhaled or topical, are not permitted within 3 months prior to Visit 1 or during the study
* Current and/or previous use of finasteride (Proscar, Propecia) or dutasteride (GI198745, AVODART™) exposure within 6 months prior to Visit 1
* Anabolic steroids within 6 months prior to Visit 1
* Participation in any other investigational or marketed drug trial within the 30 days prior to Visit 1 or any time during the study period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (58):
- GSK Investigational Site, Tallinn, Estonia
- Finland (3):
  - GSK Investigational Site, Kouvola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Tampere
- France (5):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Chambéry
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Orléans
- Germany (15):
  - GSK Investigational Site, Aichach, Bavaria
  - GSK Investigational Site, Hagenow, Brandenburg
  - GSK Investigational Site, Oranienburg, Brandenburg
  - GSK Investigational Site, Schwedt, Brandenburg
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Seligenstadt, Hesse
  - GSK Investigational Site, Leer, Lower Saxony
  - GSK Investigational Site, Wismar, Mecklenburg-Vorpommern
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Dessau, Saxony-Anhalt
  - GSK Investigational Site, Eisleben Lutherstadt, Saxony-Anhalt
  - GSK Investigational Site, Hettstedt, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Ilmenau, Thuringia
- Netherlands (7):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Tilburg
  - GSK Investigational Site, Winterswijk
- GSK Investigational Site, Moscow, Russia
- Spain (15):
  - GSK Investigational Site, Alava
  - GSK Investigational Site, Alcala de Henares (madrid)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bormujo (sevilla)
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Mendaro, Guipuzcoa
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
- Sweden (5):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Uppsala
- United Kingdom (6):
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Stevenage, Hertfordshire
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, High Heaton, Newcastle Upon Tyne

REFERENCES:
- [Derived] Schroder F, Bangma C, Angulo JC, Alcaraz A, Colombel M, McNicholas T, Tammela TL, Nandy I, Castro R. Dutasteride treatment over 2 years delays prostate-specific antigen progression in patients with biochemical failure after radical therapy for prostate cancer: results from the randomised, placebo-controlled Avodart After Radical Therapy for Prostate Cancer Study (ARTS). Eur Urol. 2013 May;63(5):779-87. doi: 10.1016/j.eururo.2012.11.006. Epub 2012 Nov 12. PMID 23176897

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral dose of 0.5 milligrams (mg) matching placebo capsule once daily for 2 years
- Dutasteride 0.5 mg: Oral dose of 0.5 mg dutasteride capsule once daily for 2 years
Period: Overall Study
Arm/Group | Placebo | Dutasteride 0.5 mg
Started | 147 | 147
Completed | 76 | 111
Not Completed | 71 | 36
Not completed — Physician Decision | 18 | 4
Not completed — Withdrawal by Subject | 11 | 4
Not completed — Adverse Event | 5 | 5
Not completed — Lack of Efficacy | 2 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Met Protocol-defined Stopping Criteria | 32 | 16
Not completed — Randomized in Error | 1 | 2
Not completed — Hospitalized; Unable to Continue | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dutasteride 0.5 mg | Total
Number analyzed (Participants) | 147 | 147 | 294
Age Continuous [Mean (Standard Deviation); unit: Years] | 68.6 (6.53) | 69.7 (5.76) | 69.1 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 147 | 147 | 294
Race/Ethnicity, Customized [Number; unit: participants]
  White - Caucasian/European Heritage | 145 | 147 | 292
  White - Arabic/North African Heritage | 1 | 0 | 1
  Asian - Central/Soth Asian Heritage | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Prostate-specific Antigen (PSA) Doubling From Baseline (in Days)
Description: Time to PSA doubling is defined as the number of days between the baseline date and the study day of the first post-baseline PSA evaluation date (within treatment period, typically up to 24-month evaluations) on which the PSA value was at least twice as much as the baseline PSA value, and the immediate subsequent value, if available, was at least 85% of two times the baseline value. Participants who never achieved PSA doubling were censored at the last post-baseline, non-missing PSA evaluation.
Time Frame: up to 28 months
Population: ITT Population: all participants randomized to study treatment. Participants not having any post-baseline PSA measurements could not be evaluated and were hence excluded from this analysis (3 in placebo arm; 1 in dutasteride arm). Only participants who experienced PSA doubling (82 in placebo, 41 in dutasteride) contributed to summary statistics.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
days
  Participants (par.) with PSA doubling; n=82, 41 | 365.5 [90 to 736] | 458.0 [91 to 736]
  Par. without PSA doubling (censored); n=62, 105 | NA [NA to NA] — Data were not summarized for participants with censored time. | NA [NA to NA] — Data were not summarized for participants with censored time.
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.001, Log Rank — Comparing 24-month survival curves (includes time to PSA doubling as well as time to censoring); stratified by site cluster and previous therapy; Relative Risk (Hazard Ratio) = 0.34, 95% CI 2-sided [0.23 to 0.50] — Relative risk of dutasteride compared to placebo, derived from Cox Proportional Hazard model stratified by site cluster and previous therapy

2. Secondary Outcome: Time to Disease Progression From Baseline (in Days)
Description: Time to disease progression is defined as the number of days between baseline and the first occurrence of any of the following: PSA doubling time (PSADT)<=91 days, PSA value is at least 50% more than baseline value (>20 nanogram/milliliter [ng/ml] for primary radiotherapy group or >10 ng/ml for radical prostatectomy group), rescue treatment, cancer-positive biopsy, cancer-positive bone scan. (Confirmation of PSA criteria is required in an immediate subsequent PSA, if available, and PSA values for consideration are restricted to treatment period, typically up to 24-month evaluations.)
Time Frame: up to 28 months
Population: ITT Population. Only those participants with disease progression have been summarized.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 49 | 25
days | 365.0 [39 to 824] | 285.0 [22 to 808]

3. Secondary Outcome: Number of Participants With Disease Progression
Description: Disease progression is defined as the first occurrence of any of the following: PSADT<=91 days, PSA value is at least 50% more than baseline value (>20 ng/ml for primary radiotherapy group or >10 ng/ml for radical prostatectomy group), rescue treatment, cancer-positive biopsy, cancer-positive bone scan. If one of the PSA criteria is qualifying (within treatment period, typically up to 24-month evaluations), an immediate subsequent PSA, if available, must confirm either criterion (or at least 85% of the qualifying value).
Time Frame: up to 28 months
Population: ITT Population. Participants not having any post-baseline PSA measurements could not be evaluated and were hence excluded from this analysis (3 in placebo arm, 1 in dutasteride arm).
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
participants
  With disease progression | 49 | 25
  Without disease progression | 95 | 121

4. Secondary Outcome: Number of Participants Classified as Treatment Responders at Months 3, 6, 9, 12, 15, 18, 21, and 24
Description: Treatment responders at Month X were defined as participants (par.) with either a PSA decrease or an increase <=15% from baseline to Month X confirmed in all PSA measurements between baseline (BL) and Month X.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: ITT Population. Par. not having a post-BL measurement could not be evaluated and were hence excluded from this analysis (3 in placebo arm, 1 in dutasteride arm). Different par. may contribute data at different time points (TP); the number of par. analyzed at each TP are those with BL as well as post-baseline data at the particular TP.
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
participants
  Month 3, n=141, 141 | 64 | 117
  Month 6, n=131, 135 | 36 | 105
  Month 9, n=121, 129 | 22 | 95
  Month 12, n=110, 124 | 13 | 87
  Month 15, n=100, 121 | 10 | 82
  Month 18, n=95, 120 | 8 | 76
  Month 21, n=83, 112 | 7 | 70
  Month 24, n=76, 110 | 6 | 62

5. Secondary Outcome: Time to PSA Rise From Baseline (in Days)
Description: A participant was designated as having a PSA rise if there existed a post-baseline PSA value (within treatment period, typically up to 24-month evaluations) that was >1.15 times the baseline PSA value, and all subsequent PSA values were >1.15 times the baseline PSA value. The study day for the first PSA evaluation that qualified for analysis of PSA rise was used for time to PSA rise. If none of the post-baseline PSA values qualified for analysis of PSA rise during the study, time to PSA rise was censored at the last post-baseline PSA evaluation.
Time Frame: up to 28 months
Population: ITT Population. Only those participants with PSA rise have been summarized.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 127 | 72
days | 100.0 [39 to 729] | 279.0 [22 to 805]

6. Secondary Outcome: Number of Participants With a PSA Rise From Baseline
Description: A participant was designated as having a PSA rise if there existed a post-baseline PSA value (within treatment period, typically up to 24-month evluations) that was >1.15 times the baseline PSA value, and all subsequent PSA values were >1.15 times the baseline PSA value.
Time Frame: up to 28 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
participants
  With PSA rise | 127 | 72
  Without PSA rise | 17 | 74

7. Secondary Outcome: Time to PSA Progression (in Days)
Description: A participant was designated as having PSA progression if there existed a post-baseline PSA value (within treatment period, typically up to 24-month evaluations) that was >10 ng/ml if radical prostatectomy or >20 ng/ml if primary radiotherapy and PSA >=1.5 times the baseline PSA value, or 0<PSADT<=91 days, and all subsequent PSA values satisfied these criteria. The study day for the first PSA qualifying for progression was used for time to PSA progression. If none of the PSA values qualified for PSA progression, time to PSA progression was censored at the last post-baseline PSA evaluation.
Time Frame: up to 28 months
Population: ITT Population. Only those participants with PSA progression have been summarized.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 25 | 19
days | 368.0 [90 to 736] | 368.0 [22 to 735]

8. Secondary Outcome: Number of Participants With PSA Progression
Description: A participant was designated as having a PSA progression if there existed a post-baseline PSA value (within treatment period, typically up to 24-month evaluations) that was (>10 ng/ml if radical prostatectomy or >20 ng/ml if primary radiotherapy) and PSA >=1.5 times the baseline PSA value), or 0<PSADT<=91 days, and all subsequent PSA values satisfied either of these criteria.
Time Frame: up to 28 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
participants
  With PSA progression | 25 | 19
  Without PSA progression | 119 | 127

9. Secondary Outcome: Change in Total PSA From Baseline at Months 12 and 24
Description: Change in PSA from baseline at Month X = Month X PSA - Baseline PSA. The missing PSA value for scheduled visits could have been replaced by non-missing PSA values within 30 days after the clinic visit date. If such replacement was not possible, the latest non-missing post-baseline PSA before the scheduled visit was used for the scheduled visit PSA (Last Observation Carried Forward).
Time Frame: Baseline; Months 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/ml)
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
nanograms/milliliter (ng/ml)
  Month 12 | 2.3 (4.86) | 0.9 (7.25)
  Month 24 | 3.9 (6.09) | 2.3 (7.60)

10. Secondary Outcome: Percent Change in Total PSA From Baseline at Months 12 and 24
Description: Percent change in PSA from baseline at Month X = 100*(Month X PSA - Baseline PSA)/Baseline PSA. The missing PSA value for scheduled visits could have been replaced by non-missing PSA values within 30 days after the clinic visit date. If such replacement was not possible, the latest non-missing post-baseline PSA before the scheduled visit was used for the scheduled visit PSA (Last Observation Carried Forward).
Time Frame: Baseline; Months 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
percent change
  Month 12 | 93.1 (115.02) | 11.8 (103.41)
  Month 24 | 197.3 (282.41) | 86.2 (193.95)

11. Primary Outcome: Number of Participants With PSA Doubling From Baseline
Description: PSA doubling is defined as the first post-baseline PSA value (within treatment period, typically up to 24-month evaluations) that was at least twice as much as the baseline PSA value and was confirmed as such (at least 85% of two times the baseline PSA value) in the immediate subsequent PSA value if one is available.
Time Frame: up to 28 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
participants
  With PSA doubling | 82 | 41
  Without PSA doubling | 62 | 105
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.001, Mantel-Haenszel Chi-Square — Comparing percentages of participants with PSA doubling: 57% versus 28%

12. Primary Outcome: Time to PSA Doubling From Baseline (in Days) Within Year 1
Description: Time to PSA doubling is defined as the number of days between the baseline date and the study day of the first post-baseline PSA evaluation date within Year 1 (Y1; within treatment period, typically up to 12-month evaluations) on which the PSA value was at least twice as much as the baseline PSA value, and the immediate subsequent value, if available, was at least 85% of two times the baseline value.
Time Frame: up to 16 months
Population: ITT Population. Participants not having any post-baseline PSA measurements could not be evaluated and were hence excluded from this analysis (3 in placebo arm, 1 in dutasteride arm). Only participants with PSA doubling within Year 1 (50 in placebo, 15 in dutasteride) contributed to summary statistics.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
days
  Participants with PSA doubling in Y1; n=50, 15 | 273.5 [90 to 486] | 183.0 [91 to 383]
  Participants without PSA doubling in Y1: n=94, 131 | NA [NA to NA] — Data were not summarized for participants with censored time. | NA [NA to NA] — Data were not summarized for participants with censored time.
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.001, Log Rank — Comparing 12-month survival curves (includes time to PSA doubling as well as time to censoring); stratified by site cluster and previous therapy; Relative Risk (Hazard Ratio) = 0.25, 95% CI [0.14 to 0.45] — [estimate comment as in outcome 1, analysis 1]

13. Primary Outcome: Number of Participants With PSA Doubling From Baseline During Year 1
Description: PSA doubling is defined as the first post-baseline PSA value (within treatment period, typically up to 12-month evaluations) that was at least twice as much as the baseline PSA value and was confirmed as such (at least 85% of two times the baseline PSA value) in the immediate subsequent PSA value if one is available.
Time Frame: up to 16 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
participants
  With PSA doubling | 50 | 15
  Without PSA doubling | 94 | 131
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.001, Mantel-Haenszel Chi-Square — Comparing percentages of participants with PSA doubling: 35% versus 10%

14. Secondary Outcome: Change in PSA From Nadir PSA at Months 12 and 24
Description: Change from nadir PSA at Month X = Month X PSA - nadir PSA. Nadir PSA was reported by the site as the lowest historical PSA value after the radical therapy. A nadir value below the detection level was captured as 0.0. The missing PSA value for scheduled visits could have been replaced by non-missing PSA values within 30 days after the clinic visit date. If such replacement was not possible, the latest non-missing post-baseline PSA before the scheduled visit was used for the scheduled visit PSA (Last Observation Carried Forward).
Time Frame: Baseline; Months 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 146
ng/ml
  Month 12 | 4.7 (6.31) | 3.5 (9.04)
  Month 24 | 6.3 (7.34) | 4.9 (9.65)

15. Secondary Outcome: Percent Change in PSA From Nadir PSA at Months 12 and 24
Description: Percent change from nadir PSA at Month X = 100*(Month X PSA - nadir PSA)/Nadir PSA. Nadir PSA was reported by the site as the lowest historical PSA value after the radical therapy. A nadir value below the detection level was captured as 0.0. The missing PSA value for scheduled visits could have been replaced by non-missing PSA values within 30 days after the clinic visit date. If such replacement was not possible, the latest non-missing post-baseline PSA before the scheduled visit was used for the scheduled visit PSA (Last Observation Carried Forward).
Time Frame: Baseline; Months 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 94 | 98
percent change
  Month 12 | 2810.3 (4062.48) | 2120.7 (5284.72)
  Month 24 | 4036.1 (5860.98) | 2927.2 (6146.34)

16. Secondary Outcome: Number of Participants With the Indicated Change in PSA Doubling Time (PSADT) From Baseline at Month 12, Month 24, and End-of-treatment (up to 28 Months)
Description: Participants with improvement included those whose PSADT at a specified visit was positive but more than the baseline PSADT, whose PSA at the visit was the same as the baseline PSA, or whose PSA at the visit was less than the baseline PSA. Participants with worsening included those whose PSADT at the visit was positive but less than the baseline PSADT.
Time Frame: Baseline; Month 12, Month 24, End-of-Treatment (up to 28 months)
Population: ITT Population. Participants having no baseline (BL) PSADT (due to incomplete PSA data or no rise in PSA at BL) or no post-BL measurement could not be evaluated and were hence excluded from this analysis (3 in placebo arm, 3 in dutasteride arm). Participants with missing PSA data at a specific visit were excluded from that visit's analysis .
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 144
participants
  Month 12, Worsening; n=110, 123 | 20 | 7
  Month 12, No change; n=110, 123 | 0 | 0
  Month 12, Improvement; n=110, 123 | 90 | 116
  Month 24, Worsening; n=76, 110 | 7 | 3
  Month 24, No change; n=76, 110 | 0 | 0
  Month 24, Improvement; n=76, 110 | 69 | 107
  End-of treatment, Worsening; n=144, 144 | 37 | 19
  End-of treatment, No change; n=144, 144 | 0 | 0
  End-of treatment, Improvement; n=144, 144 | 107 | 125

17. Secondary Outcome: Changes From Baseline in Disease-related Anxiety Measured by the Memorial Anxiety Scale for Prostate Cancer (MAX-PC)
Description: MAX-PC is an 18-item, self-reported measure that evaluates prostate cancer-related anxiety. The score ranges from 0 to 54, and an increase in the score indicates a worsened anxiety level. Change from Baseline at Month X = Month X MAX-PC score - Baseline MAX-PC score. A missing post-baseline value is replaced by the last available post-baseline value (Last Observation Carried Forward(LOCF)). A general linear model controls for previous therapy, site cluster, and baseline MAX-PC score.
Time Frame: Baseline; Months 3, 6, 12, 18, and 24
Population: ITT Population. Participants not having a baseline value or not having any post-baseline value could not be evaluated for this endpoint and were hence excluded from this analysis (3 in placebo arm, 4 in dutasteride arm). Participants were excluded from a specific visit analysis if the value for the visit (after LOCF application) was missing.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 144 | 143
scores on a scale
  Month 3, n=144, 141 | -1.6 (0.63) | -1.4 (0.63)
  Month 6, n=144, 143 | -2.2 (0.63) | -3.1 (0.62)
  Month 12, n=144, 143 | -0.8 (0.72) | -2.9 (0.72)
  Month 18, n=144, 143 | -1.1 (0.79) | -2.2 (0.78)
  Month 24, n=144, 143 | -0.4 (0.78) | -1.4 (0.77)

18. Secondary Outcome: Number of Participants With a Shift From Normal at Baseline to at Least One Abnormal Laboratory Value for Any Parameter Any Time During the Study
Description: A participant has a normal value for a laboratory parameter if the value is within the low and high range of normal provided by the laboratory. Each laboratory parameter is evaluated for shift from normal at baseline to abnormal any time post-baseline. A participant with any laboratory parameter showing this shift is counted. A participant is counted only once even if he had such a shift in more than one laboratory parameter or more than once among all post-baseline evaluations.
Time Frame: Baseline; up to 28 months
Population: ITT Population. Participants not having any baseline measurements, or having a baseline but no post-baseline measurements of at least one of the same parameter could not be evaluated and were hence excluded from this analysis (7 in placebo arm, 9 in dutasteride arm).
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 140 | 138
participants | 74 | 64

19. Secondary Outcome: Number of Participants With a Threshold Laboratory Value for Any Parameter at Baseline (BL) and Any Time Post-baseline
Description: Threshold laboratory values are defined in terms of a multiplicative factor of the testing laboratory's normal range, pre-specified in the analysis plan. A laboratory value that is above the upper limit factor multiplied by the upper limit of the normal range is considered a high threshold value. A laboratory value that is below the lower limit factor multiplied by the lower limit of the normal range is considered a low threshold value.
Time Frame: Baseline; up to 28 months
Population: ITT Population. Participants not having a baseline as well as a post-baseline measurement of at least one laboratory parameter could not be evaluated and were hence excluded from this analysis (7 in placebo arm, 9 in dutasteride arm).
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 140 | 138
participants
  Threshold at BL | 5 | 9
  Non-threshold at BL; threshold at any time post-BL | 11 | 5

20. Secondary Outcome: Number of Participants With Palpable Breast Tissue (PBT) at Baseline (BL) and Any Time Post-baseline
Description: Participants underwent clinical examination of the breasts, to evaluate for palpable breast tissue. Clinical significance of the results was determined by subjective judgment of the clinical personnel performing the examination.
Time Frame: Baseline; up to 28 months
Population: ITT Population. Only those participants with PBT at baseline or PBT at any time post-baseline were measured for clinical significance.
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 147 | 147
participants
  BL; PBT, n=147, 147 | 6 | 4
  BL; Clinically significant (CS) PBT, n=6, 4 | 0 | 0
  No BL PBT, but PBT at any time post-BL, n=147,147 | 10 | 21
  CS change in PBT; BL to any time post-BL, n=10, 21 | 0 | 4

21. Secondary Outcome: Number of Participants With Nipple Tenderness (NT) at Baseline (BL) and Any Time Post-baseline
Description: Participants underwent clinical examination of the breasts, to evaluate for nipple tenderness. Clinical significance of the results was determined by subjective judgment of the clinical personnel performing the examination.
Time Frame: Baseline; up to 28 months
Population: ITT Population. Only those participants with NT at baseline or NT at any time post-baseline were measured for clinical significance.
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 147 | 147
participants
  BL; NT, n=147, 147 | 0 | 3
  BL; Clinically significant (CS) NT, n=0, 3 | 0 | 0
  No NT at BL, but NT at any time post-BL, n=147,147 | 8 | 11
  CS change in NT; BL to any time post-BL, n=8, 11 | 0 | 1

22. Secondary Outcome: Number of Participants With a Digital Rectal Examination (DRE) Evaluation Changing From Normal/Diffusely Enlarged at Baseline to Focal Abnormality at Any Time Post-baseline
Description: Participants underwent a digital rectal examination to evaluate for focal abnormality of the prostate.
Time Frame: Baseline; up to 28 months
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 147 | 147
participants | 10 | 8

23. Secondary Outcome: Number of Participants With Threshold Vital Signs at Baseline and Any Time Post-baseline
Description: Threshold vital signs are defined as follows: < 80 mmHg or > 165 mmHg for systolic blood pressure; < 40 mmHg or > 105 mm Hg for diastolic blood pressure, < 40 beats per minute (bpm) or > 100 bpm for heart rate.
Time Frame: Baseline; up to 28 months
Population: ITT Population. Participants not having a baseline as well as a post-baseline measurement of at least one vital sign parameter were excluded from this analysis (6 in placebo arm, 4 in dutasteride arm).
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 141 | 143
participants
  Baseline | 18 | 15
  Any time post-baseline | 37 | 36

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from Baseline to the End of Study (up to 28 months after treatment start).
Description: All safety analyses were performed using the ITT Population.
Arm/Group | Placebo | Dutasteride 0.5 mg
Serious Adverse Events (participants affected / at risk) | 16/147 | 16/147
Other Adverse Events (participants affected / at risk) | 31/147 | 32/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | Dutasteride 0.5 mg (N=147)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Urethral abscess (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder neck sclerosis (Renal and urinary disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | Dutasteride 0.5 mg (N=147)
Nasopharyngitis (Infections and infestations) | 10 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 4
Gynaecomastia (Reproductive system and breast disorders) | 4 | 10
Hypertension (Vascular disorders) | 10 | 4
Urinary incontinence (Renal and urinary disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.